CLINICAL TRIAL: NCT03480256
Title: Phase Id Trial to Evaluate SHR6390 Combined With Pyrotinib in Patients With HER2 Positive Advanced Stage Gastric Carcinoma
Brief Title: Study to Evaluate SHR6390 Combined With Pyrotinib in Patients With HER2 Positive Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Head of Department of Gastrointestinal Oncology,Peking University Cancer Hospital, Peking University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR6390-Id
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
Keywords: SHR6390; Pyrotinib; gastric cancer; Her-2 positive
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR6390 combined with pyrotinib (Experimental): Group A:pyrotinib 400mg qd combined with SHR 6390 100mg qd Group B: pyrotinib 400mg qd combined with SHR 6390 125mg qd Group C: pyrotinib 400mg qd combined with SHR 6390 150mg qd Group D: pyrotinib 400mg qd combined with SHR 6390 175mg qd Group E: pyrotinib 320mg qd combined with SHR 6390 100mg qd
  Interventions: Drug: SHR6390

INTERVENTIONS:
Drug: SHR6390 — SHR6390 is a novel small molecule inhibitor specifically targeting the CDK4/6 pathway.Pyrotinib is an irreversible pan-ErbB inhibitor which shows promising antitumour activity in patients with HER2-positive metastatic gastric cancer

SUMMARY:
The aim of the study is to assess the safety and tolerability of SHR6390 combined with pyrotinib in the patients with Her-2 positive advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients definitely diagnosed by pathology as Her2 positive stage III/IV gastric cancer
* 18-75 years old, ECOG PS:0-1,Life expectancy of more than12 weeks;
* Patients treated with systematic treatment to metastatic disease then experienced progressive disease
* Patients with at least one evaluable or measurable disease per RECIST v1.1
* Main organs function is normal;
* Patients should be voluntary and sign the informed consent before taking part in the study;

Exclusion Criteria:

* • Patients who have uncontrollable effusion with clinical symptoms such as severe pleural effusion and peritoneal effusion;

  * A variety of factors that affect oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea, intestinal obstruction, etc.)
  * Patients who have steroid treatment for more than 30 days or need long-term steroid treatment;
  * Patients who had previously received chemotherapy，radiotherapy, hormonotherapy,surgery,targeted therapy(including Trastuzumab) within 2 weeks ;patients who had previously received nitrosourea or Mitomycin with 6 weeks;
  * Previous treatment-related adverse events did not recover to less than 2 levels except hair loss or other conditions that did not affect the enrollment according to investigators;
  * Patients who have participated in other anticancer drug clinical trials within 4 weeks except that trial is observational or at follow up stage;
  * Patients who have uncontrollable hypomagnesemia or hypokalemia;
  * Patients with untreated or symptomatic brain metastasis;
  * Patients with malignant tumors within 5 years, except for basal cell carcinoma,squamous skin cancer and cervical carcinoma in situ;
  * Patients who are being treated with any other anticancer strategies;
  * Patients with allergic constitution or being allergic to any element in the study drugs;
  * Patients with definite gastrointestinal bleeding tendency, including: active ulcer lesions with OB(++);melena or haematemesis history within 2 months; patients with OB(+) but without tumor resection need gastroscopy. If there is active bleeding, it's not suitable for this trial;
  * Patients with active infection, including tuberculosis;
  * Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history;
  * Patients who have had severe cardiac disease within six months, including acute coronary syndrome, arrhythmias that require medication or with clinical significance, or need continuous medication that may cause QT extension, acute myocardial infarction,heart failure,and any other condition that is not suitable for this experiment according to the investigators;
  * Patients who are pregnant or breast feeding;
  * Patients who don't agree on contraception; Patients with concomitant diseases which could seriously endanger themselves or those who won't complete the study according to investigators such as hypertension, severe diabetes and thyroid diseases;
  * Patients with bad addiction such as excessive drinking or smoking;
  * Patients with definite mental disorder, including epilepsy and dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 42 days

SECONDARY OUTCOMES:
Maximum Plasma Concentration | 42 days
Area Under the Curve | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Department of GI Oncology, Peking University Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Z, Xu Y, Gong J, Kou F, Zhang M, Tian T, Zhang X, Zhang C, Li J, Li Z, Lai Y, Zou J, Zhu X, Gao J, Shen L. Pyrotinib combined with CDK4/6 inhibitor in HER2-positive metastatic gastric cancer: A promising strategy from AVATAR mouse to patients. Clin Transl Med. 2020 Aug;10(4):e148. doi: 10.1002/ctm2.148. PMID 32898333